CLINICAL TRIAL: NCT01569373
Title: Analysis of Biomarkers for Acute Graft-versus-Host Disease (GVHD).
Status: Withdrawn | Type: Observational
Why Stopped: Resources needed to complete the study were not able to be obtained.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark R. Litzow, MD, Mayo Clinic
Other Study IDs: 12-001493
Record Dates: First submitted 2012-03-29; First posted 2012-04-03 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Blood Stem Cell Transplant Failure
Keywords: Allogeneic stem cell transplant; Graft versus Host Disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post allogeneic SCT patients: Patients who have undergone an allogeneic stem cell transplant.

SUMMARY:
Samples of blood and urine will be analyzed for biomarkers to check their predictivity of Graft-versus-Host Disease (GVHD) outcomes.

DETAILED DESCRIPTION:
To determine if serum biomarkers of inflammation correlate with onset and severity of acute GVHD, particularly GVHD of the gut.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older patients
* Undergoing allogeneic stem cell transplant

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone an allogeneic stem cell transplant being followed for post transplant care.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of severe acute GVHD | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Litzow, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States